CLINICAL TRIAL: NCT07355582
Title: Injury Incidence, Severity and Burden Over Two Consecutive Seasons in French Elite Youth Rugby Players of Rugby Club Toulonnais
Brief Title: Injury Incidence, Severity and Burden in Elite Youth Rugby Players
Acronym: RUBYS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Rugby Club Toulonnais Association (Unknown); Rugby Club Toulonnais S.A.S.P (Unknown); Laboratoire Jeunesse - Activité Physique et Sportive - Santé (J-AP2S), Université de Toulon (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-016
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rugby-related Injuries
Keywords: Injury; Sport Injury; Sport prevention; Rugby; Injury incidence
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- French elite youth rugby players of Rugby Club Toulonnais: Youth rugby players (boys and girls, aged 13-18) licensed in RCT Association elite youth program (U14, U15, U16, U18) who present at least one injury during the two-season study period. Medically followed by the Sports Medicine and Traumatology Unit (UMTS).
  Interventions: Other: Medical consultation

INTERVENTIONS:
Other: Medical consultation — Injury-related medical consultations provided by the Sports Medicine and Traumatology Unit (UMTS) at Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer (CHITS)

SUMMARY:
Observational cohort study, with a closed, both retrospective and prospective design, aiming to describe the incidence, severity, and burden of injuries among male and female players enrolled in the Rugby Club Toulonnais (RCT) Association program (U14 to U18 categories) over two consecutive seasons (2024-2025 and 2025-2026), based on routinely collected medical data recorded in the Askamon software.

Youth male and female players registered with the RCT Association program, starting from the U14 category, and enrolled in partner school structures within the Toulon Metropolitan area. These players benefit from an integrated academic and athletic support program.

Inclusion criteria: male or female players licensed with the RCT Association from the U14 category and above; under the medical supervision of the RCT Association; having sustained at least one injury requiring a medical consultation between August 1, 2024, and June 30, 2026; non-opposition from the participant and/or their legal guardians after being informed about the study.

Exclusion criteria: opposition from the participant or their parents/legal guardians to the use of personal data for research purposes; players not under the medical responsibility of the RCT Association.

Enrollment (estimated): approximately 200 licensed players per season, with an estimated 400 injuries per season, and exhaustive inclusion of all injured players from the active registry over two seasons.

DETAILED DESCRIPTION:
The RUBYS study is an observational closed cohort conducted over two consecutive competitive seasons (2024-2025 and 2025-2026) in youth rugby players from the RCT (Rugby Club Toulonnais) Association. It focuses on the epidemiology of rugby-related injuries in adolescents enrolled in a structured dual project (school and sport) in the Toulon metropolitan area.

Young players (boys and girls) aged approximately 13 to 18 years, licensed in the RCT Association from the U14 category upwards, benefit from adapted school timetables and regular supervised training sessions. These athletes are monitored medically by the Sports Medicine and Traumatology Unit (UMTS) of the Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer (CHITS), under the responsibility of the principal investigator. All injuries requiring medical consultation are routinely recorded in the Askamon software, which centralizes clinical information, exposure data and follow-up for each player.

The study does not modify usual care and does not introduce any additional medical procedures beyond those required for standard injury management. When an injury occurs, the player is assessed and treated according to usual practice (club doctor, attending physician or emergency services, with referral to specialists and use of imaging or surgery if needed). Information regarding the type of injury, anatomical location, circumstances, and days lost from rugby is recorded as part of routine clinical documentation and sports records (match sheets, training attendance registers), then entered into Askamon. No specific intervention, randomization or additional biological sampling is planned within the framework of this protocol.

For the purposes of the study, a pseudonymized extraction of Askamon will be performed and will include all players with at least one injury requiring medical consultation between August 1, 2024, and June 30, 2026. Each injury event will be considered as an observation, and multiple injuries in the same player will be analysed separately. The dataset will include demographic variables (age, sex), relevant medical history where available, detailed injury characteristics (diagnosis, lesion type, involved body region) and severity expressed as time-loss days until full return to competition. Injuries will be categorized according to international rugby consensus definitions (World Rugby/International Rugby Board [IRB]) to ensure comparability with existing literature.

Non-medical variables related to rugby participation will also be extracted: playing position (forwards or backs), competition category, context of occurrence (match versus training), match situation or training drill, recurrence, playing surface (natural or synthetic), type of competition, venue, period of the season, environmental conditions (temperature, weather), equipment (footwear condition) and perceived fatigue where available. These contextual factors will be used to explore potential modifiable risk factors and high-risk situations. The exposure denominator (player-hours) will be estimated from training and match schedules, attendance records and competition data provided by the RCT Association.

The primary analysis will consist of calculating injury incidence rates expressed as the number of injuries per 1000 player-hours of exposure, overall and stratified by sex, age category, playing position and context (training versus match). Secondary analyses will describe the distribution of injuries by type, anatomical site and severity categories, and will assess the relative contribution of different mechanisms and contexts to overall injury burden. Time-loss injuries will be classified into predefined severity grades based on the number of days of absence from full rugby participation, allowing the identification of injuries with the highest impact on players and on team performance.

From a methodological standpoint, the study is primarily descriptive, aiming at providing precise estimates of incidence and severity in the entire eligible population, rather than testing a specific intervention. All eligible players will be included, so no formal a priori sample size calculation is required. The precision of incidence estimates (95% confidence intervals) will be evaluated post hoc according to the actual number of injuries and exposure hours collected. Where appropriate, multivariable models may be used to explore associations between injury occurrence and potential risk factors (e.g. position, age category, match versus training, playing surface), while acknowledging the observational nature of the data and the limitations regarding causal inference.

Participants and their legal guardians will be informed through a written information letter describing the objectives of the research, the nature of the data used, the pseudonymization process and their rights (access, rectification, opposition and withdrawal). Non-opposition from parents or legal guardians is required for inclusion. In case of withdrawal, all data relating to the concerned player will be definitively deleted from the research dataset. No additional burden or constraint is imposed on players, families or staff.

Data will be pseudonymized before analysis, with the identification key kept securely at the Sports Medicine and Traumatology Unit (UMTS) of the CHITS and not available to the statisticians. The dataset will be stored on secure institutional servers, in compliance with applicable regulations on personal data protection. Data will be retained for a limited period (up to 2 years after the last publication, or 3 years after the end of data collection in the absence of publication), then archived for 15 years according to national regulations on clinical research archiving. Results will be disseminated through scientific publications and presentations, with the aim of informing prevention strategies, improving rehabilitation pathways and contributing to safer rugby practice in youth populations.

ELIGIBILITY:
Inclusion Criteria:

* Licensed players (boys or girls) in the RCT Association program from U14 category onwards
* Players presenting at least one injury requiring medical consultation between 01/08/2024 and 30/06/2026

Exclusion Criteria:

* Opposition from participant or parents to participate in the research
* Players not under medical responsibility of the RCT Association

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth rugby players (boys and girls, aged 13-18) licensed in RCT Association elite youth program (U14, U15, U16, U18). Integrated in specialized schools of Toulon metropolitan area with adapted schedules for dual academic-sport pathway. Medically followed by the Sports Medicine and Traumatology Unit (UMTS) at Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer (CHITS). All injuries recorded in Askamon database.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Injury incidence rate among youth rugby players over two consecutive seasons | Up to 24 months
  Number of injuries requiring a medical consultation divided by the total number of player-hours of exposure (training and matches), expressed as injuries per 1000 player-hours.

SECONDARY OUTCOMES:
Distribution of injuries by type and anatomical location. | Up to 24 months
  Proportion of injuries categorized by pathological category (e.g. sprain, fracture, contusion, concussion) and by anatomical region (e.g. upper limb, lower limb, head/neck, trunk).
Context of injury occurrence (match versus training, playing position and competition category). | Up to 24 months
  Proportion of injuries occurring in matches versus training sessions, and distribution of injuries according to playing position (forwards or backs) and player category (U14, U15, U16, U18).
Frequency of recurrent injuries. | Up to 24 months
  Number and proportion of players sustaining more than one injury during the two-season study period, and number of recurrent injuries per player.
Injury severity according to time-loss days. | Up to 24 months
  Distribution of injuries by severity grade: Grade 0 (no time loss), Grade 1 (1-3 days), Grade 2 (4-7 days), Grade 3 (8-28 days), Grade 4 (>28 days).
Injury mechanisms. | Up to 24 months
  Distribution of injuries by mechanism (running, tackling, ruck)
Environmental factors. | Up to 24 months
  Distribution of injuries by environmental factors (playing surface, weather conditions, equipment status, and fatigue state).
Level of care. | Up to 24 months
  Injury management will be detailed by level of care (on-field and off-field).
Medical specialist referrals. | Up to 24 months
  Injury management will be detailed by medical specialist referrals.
Use of diagnostic facilities. | Up to 24 months
  Injury management will be detailed by use of diagnostic facilities.
Medical procedures. | Up to 24 months
  Injury management will be detailed by treatment or surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan CANESSA, Strength/conditioning coach, Study Director — RCT Association; Jean-Jacques RAYMOND, MD, Principal Investigator — CHITS
Locations (2):
- France (2):
  - CHITS, Toulon, Var
  - RCT Association, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A King D, N Clark T, A Hume P, Hind K. Match and training injury incidence in rugby league: A systematic review, pooled analysis, and update on published studies. Sports Med Health Sci. 2022 Mar 27;4(2):75-84. doi: 10.1016/j.smhs.2022.03.002. eCollection 2022 Jun. PMID 35782281
- [Background] Cruz-Ferreira A, Cruz-Ferreira E, Santiago L, Taborda Barata L. Epidemiology of injuries in senior male rugby union sevens: a systematic review. Phys Sportsmed. 2017 Feb;45(1):41-48. doi: 10.1080/00913847.2017.1248224. Epub 2016 Oct 26. PMID 27741401
- [Background] Leahy TM, Kenny IC, Campbell MJ, Warrington GD, Cahalan R, Harrison AJ, Lyons M, Glynn LG, Comyns TM. Injury surveillance in school Rugby: A systematic review of injury epidemiology & surveillance practices. Phys Ther Sport. 2019 Jul;38:170-178. doi: 10.1016/j.ptsp.2019.05.005. Epub 2019 May 25. No abstract available. PMID 31158741
- [Background] Fuller CW, Molloy MG, Bagate C, Bahr R, Brooks JH, Donson H, Kemp SP, McCrory P, McIntosh AS, Meeuwisse WH, Quarrie KL, Raftery M, Wiley P. Consensus statement on injury definitions and data collection procedures for studies of injuries in rugby union. Br J Sports Med. 2007 May;41(5):328-31. doi: 10.1136/bjsm.2006.033282. PMID 17452684
- [Background] Thomas A, Davis K, Regnier A, López AD. Injury incidence and severity rates in male professional Rugby-15s: A systematic review. Int J Athl Ther Train. 2024. doi:10.1123/ijatt.2024-0051.